CLINICAL TRIAL: NCT02060084
Title: Effect of Early Oral Triple Viable Bifidobacterium Intestinal Flora in Preterm
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wang Hua (Industry)
Responsible Party: Sponsor-Investigator, Wang Hua, Director of pediatric, Kunshan First People's Hospital Affiliated to Jiangsu University
Organization: Kunshan First People's Hospital Affiliated to Jiangsu University (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYSD2012021
Record Dates: First submitted 2014-02-02; First posted 2014-02-11 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2014-01

CONDITIONS: Disorder of Stomach Function and Feeding Problems in Newborn; Feeding and Eating Disorders of Childhood
Keywords: preterm;; Intestinal flora;; early Micro-feeding; Feeding intolerance
MeSH Terms: conditions — Feeding and Eating Disorders of Childhood; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a control group (Experimental): a control group : the same dose of luke warm water
  Interventions: Drug: a control group
- treatment group (Experimental): treatment group: viable Bifidobacterium 0.5 bid po
  Interventions: Drug: a probiotic-supplemented group

INTERVENTIONS:
Drug: a control group — the same dose of luke warm water
  Arms: a control group
Drug: a probiotic-supplemented group — was orally administered starting from day 2 after birth, at a dose of 0.5g (the numbers of Long Bifidobacterium, Lactobacillus acidophilus and Enterococcus faecalis in live>0.5*107CFU), twice per day, for 2 weeks
  Other Names: the experimental group
  Arms: treatment group

SUMMARY:
Gut of newborn preterm is sterile, immediately by the mother and the surrounding environment from microbial colonization. As the effects of diet, intestinal flora is rapidly changed. Preterm children significantly delay in the establishment of normal flora,during hospitalization because of no breastfeeding, use of antibiotics, enteral feeding delay, combat disease and other factors. In this study, hospitalized preterm children for the study, the prospective randomized double-blind controlled study, to find oral intestinal bifidobacteria and lactobacilli and bifidobacteria subspecies composition and distribution, and further show intestinal bacteria in premature children case group.

DETAILED DESCRIPTION:
Preterm infants are at high risk of deeding intolerance especially low birth weight infants, Whether oral triple viable Bifidobacterium and early Micro-feeding may improve the symptoms of feeding intolerance.

84 preterm infants BW(birth weight) less than 2.5kg,entered neonatal intensive care unit(NICU) less than 24 hours and meet the Inclusion Criteria of this study will be Randomly divided into three groups, control group、 treatment group1 (Triple viable Bifidobacterium 0.5g bid po)、treatment group2 （Triple viable Bifidobacterium 0.5g bid po and early micro-feeding）. treatment period for more than 1 week. For three groups, feeding symptoms,the traits and frequency of stool of 3 days,1 weeks,2 weeks.And the stool flora measured by PCR.

ELIGIBILITY:
Inclusion Criteria:

* preterm with birth weight <2.5kg

Exclusion Criteria:

* Gastrointestinal bleeding and NEC,Kidney,liver function abnormal and have Serious congenital malformation

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Intestinal flora | up to one week
  measure the intestinal flora of three groups and identify the effect of early oral triple viable bifidobacterium for preterm infants

SECONDARY OUTCOMES:
Feeding intolerance | up to one week
  compare the feeding intolerance rate of three groups

CONTACTS AND LOCATIONS:
Locations (1):
- Kunshan First Hospital, Kunshan, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The patients were randomly assigned to either a control group or a probiotic-supplemented group in the following manner. The randomization schedule was made available only to the pharmacist who supervised the quality, transport and storage of LCB. Infants were followed up until they were discharged from the hospital or died. They were withdrawn from the trial if severe adverse effects developed, or parents withdrew consent. The probiotic-supplemented group were orally administered LCB (Bifico, Shanghai Xinyi Pharmaceutical Inc. Shanghai), and the control group was fed with the same dose of luke warm water); both the preparations were supplied in identical containers. LCB was orally administered starting from day 2 after birth, at a dose of 0.5g (the numbers of Long Bifidobacterium, Lactobacillus acidophilus and Enterococcus faecalis in live>0.5*107CFU), twice per day, for 2 weeks.